CLINICAL TRIAL: NCT00098826
Title: Phase I and Pharmacodynamic Study of SB-715992 in Acute Leukemias
Brief Title: SB-715992 in Treating Patients With Acute Leukemia, Chronic Myelogenous Leukemia, or Advanced Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03127; CASE 3904; U01CA062502 (NIH); U01CA062505 (NIH)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Acute Undifferentiated Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Acute Promyelocytic Leukemia (M3); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Blastic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts | interventions — ispinesib; CK0238273

ARMS (1):
- Treatment (ispinesib) (Experimental): Induction chemotherapy: Patients receive SB-715992 IV over 1 hour on days 1-3. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Consolidation chemotherapy: Patients achieving CR, PR, or SD after induction chemotherapy receive up to 4 additional courses of SB-715992 beyond CR, PR, or SD.
  Cohorts of 3-6 patients receive SB-715992 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 9 patients are treated at the MTD.
  Interventions: Drug: ispinesib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: ispinesib — Given IV
  Other Names: CK0238273; SB-715992
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of SB-715992 in treating patients who have acute leukemia, chronic myelogenous leukemia, or advanced myelodysplastic syndromes. Drugs used in chemotherapy, such as SB-715992, work in different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of SB-715992 given as a daily x 3 infusion in patients with acute leukemia.

II. To obtain pharmacokinetic studies of SB-715992 given on a 3 consecutive day schedule every 3 weeks.

III. To describe treatment-related and dose-limiting toxicities of SB-715992 in patients with acute leukemia.

IV. To describe the anti-leukemia activity of SB-715992. V. To correlate treatment-related toxicities with pharmacokinetic studies of SB-715992.

SECONDARY OBJECTIVES:

I. To validate KSP as the major target of SB-715992 by determining the impact of drug treatment on cytoskeletal morphology in peripheral blood mononuclear cells and circulating leukemic blasts.

II. To determine the expression of tubulin isoforms and KSP in leukemic blasts and explore possible relationships between gene expression and response to SB-715992.

OUTLINE: This is a dose-escalation, multicenter study.

Induction chemotherapy: Patients receive SB-715992 IV over 1 hour on days 1-3. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Consolidation chemotherapy: Patients achieving complete response (CR), partial response (PR), or stable disease (SD) after induction chemotherapy receive up to 4 additional courses of SB-715992 beyond CR, PR, or SD.

Cohorts of 3-6 patients receive SB-715992 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 9 patients are treated at the MTD.

Patients are followed for 6 weeks.

PROJECTED ACCRUAL: Approximately 15-30 patients will be accrued for this study within 7.5-15 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have acute myelogenous or acute lymphoblastic leukemia refractory to primary standard induction therapy; relapsed/refractory acute leukemia; chronic myelogenous leukemia in blast crisis are eligible at diagnosis or after failing aggressive induction chemotherapy (providing they are refractory to imatinib); acute leukemia secondary to preexisting hematologic condition or prior chemotherapy are eligible at diagnosis or after failing aggressive induction chemotherapy, advanced myelodysplastic syndrome (RAEB or RAEB-2 providing they are neutropenic or transfusion dependent); patients with de-novo acute leukemia who are not eligible for aggressive standard induction chemotherapy due to advanced age or serious comorbid medical or psychiatric conditions, patients above age 60 with de-novo AML and unfavorable cytogenetics
* At least 2 weeks must have elapsed between completion of most recent cytotoxic chemotherapy, or biologic therapy except for hydroxyurea or corticosteroids or Imatinib (24 hours); patients who have previously received an autologous stem cell transplant are allowed providing a minimum of 3 months has elapsed from transplant (T0) and patient has recovered from transplant associated toxicities; patients who have had prior allogeneic stem cell transplant are not eligible; a minimum of five days must have elapsed since administration of granulocyte or granulocyte-macrophage colony-stimulating factor and a minimum of 2 weeks if Neulasta; minimum of 2 weeks since administration of gemtuzumab, ozogamicin (Mylotarg), minimum of 4 weeks for prior investigational agents
* ECOG performance status =< 2 (Karnofsky >= 50%)
* Life expectancy of at least 4 weeks
* Direct serum bilirubin =< 1.5 mg/dl
* AST(SGOT)/ALT(SGPT) < 3 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal
* The effects of SB-715992 on the developing human fetus are unknown; for this reason and because mitotic inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not have received any other investigational agents within 28 days of study entry
* Patients may not receive any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study
* Prohibited medications: SB-715992 is a moderate to significant in vitro inhibitor of CYP3A4; the following lists of medications/substances are moderate to significant inhibitors/inducers of CYP3A4 that, if administered concomitantly with SB-715992, may alter study drug exposure; the use of these medications/substances within 14 days (>= 6 months for amiodarone) prior to the administration of the first dose of SB-715992 through discontinuation from the study is prohibited

  * Inhibitors of CYP3A4:

    * Antibiotics: clarithromycin, erythromycin, troleandomycin
    * Antifungals: itraconazole, ketoconazole, fluconazole (doses > 200 mg/day), voriconazole
    * Antidepressants: nefazodone, fluvoxamine
    * Calcium channel blockers: verapamil, diltiazem
  * Miscellaneous: amiodarone*, grapefruit juice, bitter orange; *use of amiodarone within 6 months prior to the administration of the first dose of SB-715992 is prohibited
  * Inducers of CYP3A4:

    * Anticonvulsants: phenytoin, carbamazepine, phenobarbital, oxcarbazepine
    * Antibiotics: rifampin, rifabutin, rifapentine
    * Miscellaneous: St. John's wort, modafinil
* Patients with suspected or proven CNS leukemia (diagnostic lumbar puncture not required before enrollment)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SB-715992
* Uncontrolled intercurrent illness including, but not limited to ongoing or active or poorly controlled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, poorly controlled pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with pre-existing neuropathy of grade 2 or higher are not eligible to participate
* Pregnant women are excluded from this study because SB-715992 is a mitotic inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SB-715992, breastfeeding should be discontinued if the mother is treated with SB-715992
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ispinesib, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to day 28
Pharmacokinetics of ispinesib in terms of total systemic clearance, peak concentration, area under the curve (AUC), and half-lives | Up to 96 hours post-infusion
  Summarized with histograms, medians, quartiles and ranges. Scatterplots and correlation coefficients will be used to evaluate the association between the pharmacokinetic (PK) variables and the ispinesib dose, as well the changes in the peripheral blood mononuclear cell (PBMC) values.
Treatment-related and dose-limiting toxicities of ispinesib, based on the NCI CTCAE v3.0 | Up to 2 years
Clearing of circulating peripheral blasts | By 35 days from start of most recent course of chemotherapy
Attainment of aplastic bone marrow | By 35 days from start of most recent course of chemotherapy
  Scatterplots, means, standard deviations, and confidence intervals will be constructed to compare responders and non-responders.
Achievement of complete or partial remission | By 35 days from start of most recent course of chemotherapy
  Scatterplots, means, standard deviations, and confidence intervals will be constructed to compare responders and non-responders.
Correlation between treatment-related toxicities with pharmacokinetic studies | By 35 days from start of most recent course of chemotherapy
  Scatterplots, means, standard deviations, and confidence intervals will be constructed to compare responders and non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Cooper, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States